CLINICAL TRIAL: NCT06728800
Title: Leveraging Interactive Digital Technology to Increase Access to Family-Based Behavioral Treatment for Childhood Obesity
Acronym: FBT 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: Washington University School of Medicine (Other); University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBT 2.0 DPII
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBT 2.0 (Experimental): Dyads assigned to receive FBT 2.0 will receive all eight modules over the six-month trial, completing one module every two weeks. Dyads will have free access to all completed modules for the duration of the six-month trial. Each module is expected to take approximately two to three sessions to complete, each session lasting approximately 45 minutes. At least one interventionist-led session (20-30 minutes) will occur per week, with additional sessions or coach support as needed via text exchange and/or videoconferencing supported on the website. Families will be able to engage with the software for as long as desired during the six-month trial.
  Interventions: Behavioral: FBT 2.0
- Information-and-referral Control (Other): Caregiver-youth dyads randomized to the information-and-referral control intervention will be given written educational materials. Prior to starting the intervention trial, dyads will meet for 20 minutes with a trained researcher who will provide them with educational materials used in investigators' prior studies which teaches about the impact of eating and activity behaviors on weight. Caregivers will be asked to monitor their health by using daily paper-and-pencil diaries to record eating and activity behaviors. Youth without a medical provider will be given referrals to a primary care provider in their community.
  Interventions: Behavioral: Information-and-referral

INTERVENTIONS:
Behavioral: FBT 2.0 — FBT 2.0 is a translation of Family-Based Behavioral Treatment (FBT) into an e-health intervention product for families with a child/adolescent with obesity. FBT is an evidence-based obesity intervention that takes a family-centered approach to weight management that includes training in behavioral skills for the family, such as self-monitoring, stimulus control, problem solving, pre-planning, and impulse control. Youth with obesity, along with one participating caregiver, will be introduced to the evidence- based Traﬃc Light Eating Plan and behavioral skill training appropriate for their developmental age, while the caregiver learns positive parenting approaches to help shape and support their child's weight change efforts in addition to their own weight management goals. The ﬁnal product will consist of eight modules, each aligned with evidence-based FBT skills and competencies.
  Arms: FBT 2.0
Behavioral: Information-and-referral — Caregiver-youth dyads randomized to the information-and-referral control intervention will be given written educational materials. Prior to starting the intervention trial, dyads will meet for 20 minutes with a trained researcher who will provide them with educational materials used in investigators' prior studies which teaches about the impact of eating and activity behaviors on weight. Caregivers will be asked to monitor their health by using daily paper-and-pencil diaries to record eating and activity behaviors. Youth without a medical provider will be given referrals to a primary care provider in their community.
  Arms: Information-and-referral Control

SUMMARY:
The primary goal of this SBIR Direct to Phase II is to expand upon the existing training platform to create an "all-in-one" digital product, FBT 2.0, that offers an integrated suite of intervention components, including (a) dynamic, personalized, self-paced program for children and parent/caregivers; (b) e-training and ongoing support for interventionists; and (c) family engagement and monitoring tools for interventionists. Investigators will create a comprehensive, e-learning digital intervention with engaging, interactive, and personalized online tools for youth and their parents/caregivers that are integrated into the broader interventionist platform.

DETAILED DESCRIPTION:
The primary goal of this SBIR Direct to Phase II is to expand upon the existing training platform to create an "all-in-one" digital product, FBT 2.0, that offers an integrated suite of intervention components, including (a) dynamic, personalized, self-paced program for children and parent/caregivers; (b) e-training and ongoing support for interventionists; and (c) family engagement and monitoring tools for interventionists. Investigators will create a comprehensive, e-learning digital intervention with engaging, interactive, and personalized online tools for youth and their parents/caregivers that are integrated into the broader interventionist platform. For the Pilot test , investigators will randomly assign half of the enrolled dyads (by age group i.e., 6 to 12, > 12) to FBT 2.0 and half to the information-and-referral control condition. Dyads assigned to receive FBT 2.0 will receive all eight modules over the six-month trial, completing one module every two weeks. Dyads will have free access to all completed modules for the duration of the six-month trial. Each module is expected to take approximately two to three sessions to complete, each session lasting approximately 45 minutes. At least one interventionist-led session (20-30 minutes) will occur per week, with additional sessions or coach support as needed via text exchange and/or videoconferencing supported on the website. Families will be able to engage with the software for as long as desired during the six-month trial.

Caregiver-youth dyads randomized to the information-and-referral control intervention will be given written educational materials. Prior to starting the intervention trial, dyads will meet for 20 minutes with a trained researcher who will provide them with educational materials used in investigators' prior studies which teaches about the impact of eating and activity behaviors on weight. Caregivers will be asked to monitor their health by using daily paper-and-pencil diaries to record eating and activity behaviors. Youth without a medical provider will be given referrals to a primary care provider in their community.

The same set of outcome measures will be collected for children and caregivers in both conditions at each of three timepoints: (1) prior to starting the trial (baseline); (2) at 3 months into the trial; and (3) at 6 months (after completing their last module). For all participants randomized to FBT 2.0, software usage data will be collected throughout the six-month trial and product evaluations will be collected at post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* must be youth between the ages of 6 and 18
* must have a body mass index (BMI) percentile greater than or equal to the 95th BMI percentile for age and sex
* must have one caregiver participate, who is at least 18 years of age and lives with the child at least 50% of the time.

Exclusion Criteria:

* co-morbid disorders that contraindicate weight loss (e.g., eating disorder).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Relative Weight | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  Youth: The participating caregiver is given the CDC guidelines for "Measuring Children's Height and Weight Accurately at Home." The FBT coach will review these guidelines with the caregiver to assure comprehension. Median body mass index (BMI) for that child's age (in months) and sex is based on norms defined by Kuczmarski and colleagues and available from the CDC. Percent overweight was chosen as the primary outcome measure given its sensitivity to change throughout the BMI range. Caregiver: Exploratory analyses will examine caregiver weight change, defined as percent change from weight at baseline, among caregivers who have obesity (BMI ≥ 30) at baseline.
Youth Pediatric Symptom Checklist-17 | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  Youth: The Pediatric Symptom Checklist-17 is a widely used, briefer version of the PSC-35, a caregiver-completed measure of children's psychosocial functioning, where caregivers rate each symptom on a scale of 0-2, where 0 means never, 1 means sometimes, and 2 means often.
Youth Center for Epidemiological Studies Depression Scale for Children | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  Youth: Depression is measured in children using a 20-item Center for Epidemiological Studies Depression Scale for Children. Possible scores range from 0-60 with each item response scored as 0 = Not At All, 1 = A Little, 2 = Some, and 3 = A Lot.
Caregiver Adult Patient Health Questionnaire | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  Caregiver: Adults complete the 2- item Patient Health Questionnaire to measure depression. Each symptom is scored on a scale of 0-3, with 0 = Not At All, 1 = Several Days, 2 = More than half the Days, and 3 = Nearly every day.
Family Nutrition and Physical Activity Screening Tool | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  The Family Nutrition & Physical Activity Screening Tool is a 20-item parent-report scale designed to assess family environments and practices that have been shown to be associated with children's risk of becoming overweight. Each item is scored on a 1-4 point scale with 4 representing the more favorable practice or policy.
Automated Self-Administered 24-hour Dietary Assessment Tool | Daily during 6-month trial period
  The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool is a free, web-based tool that enables automatically coded, self-administered 24-hour diet recalls that will be completed by the participating adolescent aged 13 or older, or with the caregiver's assistance (for youth < 13 years of age). The caregiver will also complete a 24-hour dietary recall for their own intake. Outcomes will be average daily kilocalories, fruit and vegetable servings, and percentage intake from fat.
Physical activity | 7 days during 6-month trial period
  Objective physical activity will be assessed for youth and caregivers using accelerometers worn on the wrist during sleep and daily activities for seven days at each assessment time point. Outcomes will be minutes of moderate or vigorous activity (physical activity) and minutes of sedentary activity.
Sizing Them Up | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  Youth: Sizing Them Up is a 22-item parent-report weight-specific quality of life measure used to assess the impact of weight on the child's health and on their day-to-day functioning. Each item is scored on a 1-4 scale, with 1 = Never, 2 = Sometimes, 3 = Often, and 4 = always, with lower scores meaning a better outcome.
Pediatric Quality of Life Inventory | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  Youth: The Pediatric Quality of Life Inventory is a modular instrument for measuring health-related quality of life in children and adolescents ages 2 to 18. Each item is scored on a scale from 0 - 4, with 0 = never a problem, 1 = almost never a problem, 2 = sometimes a problem, 3 = often a problem, and 4 = a lot of a problem, with lower scores being a more favorable outcome.
Caregiver Short Form(SF)-12 Health Survey | Baseline at start of trial, at 3-month timepoint, and at 6-month conclusion of trial
  The SF-12 Health Survey is a shorter version of the SF-36 designed to assess the caregiver's functional health and well-being, and overall quality of life. Higher scores mean a better health-related quality of life, with lower scores suggesting below-average health.
Intervention Feedback | At study completion, average of 6 months
  Caregivers and youth in both conditions will provide feedback regarding their experiences during the trial period. On a 5-point scale (1=Strongly Disagree to 5=Strongly Agree), respondents will rate the degree to which their experience was: (a) useful for increasing knowledge of weight-related behaviors; (b) useful for learning self-management skills; (c) helped with changing unhealthy behaviors; (d) valuable for families and youth with obesity; (e) engaging for families; (f) innovative compared to alternatives; and (g) better than alternatives. Additionally, child and parent satisfaction with FBT will be assessed at the end of treatment using the 8-item Client Satisfaction Questionnaire. Participants will also be asked to provide written comments, listing specific concerns or problems. Follow-up interviews via telephone by trained research assistants will be conducted to clarify responses and gather additional details, as needed.
After-Scenario Questionnaire (ASQ) | At study completion, average of 6 months
  The After-Scenario Questionnaire (ASQ) is a 3-item measure on which adolescents will rate their satisfaction with FBT 2.0.
Post-Study System Usability Questionnaire (PSSUQ) | At study completion, average of 6 months
  The Post-Study System Usability Questionnaire (PSSUQ) is a 19-item survey assessing overall user satisfaction with the system and interface.
Technology Acceptance Model (TAM) | At study completion, average of 6 months
  Technology Acceptance Model (TAM) is a 16-item measure assessing end-user acceptance of technology in the areas of perceived usefulness, perceived ease of use, and attitudes towards using.
Product Evaluation | At study completion, average of 6 months
  In addition, participants will rate (5-point scale from 1=Not at all to 5=Extremely) the quality of FBT 2.0 in the following areas: (a) user friendly; (b) easy to navigate; (c) appealing graphic design; (d) easy to follow directions; (e) jargon free; (f) engaging; (g) high quality content; (h) high value content; (i) relevance to real-life; (j) login functions; (k) search functions; and (l) help functions.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DeRosier, PhD, Principal Investigator — 3C Institute; Denise Wilfley, PhD, Principal Investigator — Washington University School of Medicine; Leonard Epstein, PhD, Principal Investigator — University at Buffalo
Locations (1):
- 3C Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated by this project will be made available upon request after the publication of the main findings from each aim. Investigators will require parties requesting data access to submit a detailed description of their plans for the data with their personal identification, institutional affiliation, a CV, estimated duration of the proposed research, source of financial support, and a conflict-of-interest statement. The MPIs will decide whether sharing of the data is appropriate or if other information and/or additional safeguards are needed. Once the request is approved, data transfer and use agreements will be developed if necessary, and the requesting investigator must obtain approval from their institution's IRB or request to rely on the IRB of record. Appropriate de- identification techniques required by both HIPAA and the Common Rule will allow for sharing of data that does not compromise participant confidentiality.